CLINICAL TRIAL: NCT06118086
Title: A Phase 1, Multicenter, Open-label Study of REM-422, a MYB mRNA Degrader, in Patients With Recurrent or Metastatic Adenoid Cystic Carcinoma
Brief Title: Study of REM-422 in Patients With Recurrent or Metastatic Adenoid Cystic Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Remix Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REM-422-101
Record Dates: First submitted 2023-10-13; First posted 2023-11-07 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Adenoid Cystic Carcinoma; Metastatic Adenoid Cystic Carcinoma; Recurrent Adenoid Cystic Carcinoma
MeSH Terms: conditions — Carcinoma, Adenoid Cystic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- REM-422 (Experimental): * Dose Escalation: Participants will receive escalating doses of REM-422 to determine Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D)-422, oral capsule administered once daily
  * Dose Expansion: Participants will receive REM-422 at the identified RP2D
  * Treatment will continue until disease progression, therapy intolerance, or participant withdrawal
  * Safety evaluation will continue until 30 days of last administration of REM-422
  Interventions: Drug: REM-422

INTERVENTIONS:
Drug: REM-422 — * REM-422 is a first in class, small molecule mRNA inhibitor that reduces expression of the MYB transcription factor
  * REM-422 will be administered orally once daily

SUMMARY:
The goal of this study is to determine the safety and antitumor effects of REM-422, a MYB mRNA degrader, in people with advanced Adenoid Cystic Carcinoma (ACC)

DETAILED DESCRIPTION:
This is a Phase 1, open-label, non-randomized, multicenter study investigating REM-422, a potent, selective, and oral small molecule mRNA degrader that reduces expression of the MYB transcription factor for patients with recurrent or metastatic ACC.

This study includes a Dose Escalation Phase and a Dose Expansion Phase. The purpose of the Dose Escalation Phase is to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of REM-422 in patients with recurrent or metastatic ACC. The purpose of Dose Expansion is to further evaluate the safety and anti-tumor activity of the RP2D carried forward from Dose Escalation.

Participation in this study will continue until disease progression, therapy intolerance, or participant withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to provide informed consent.
2. Be 18 years or older at the time of informed consent.
3. Disease criteria:

   1. Histologically confirmed ACC, any site of origin.
   2. Have locally advanced or metastatic ACC.
   3. Dose Escalation phase ONLY: Evidence of radiographic progression and/or signs and symptoms associated with their disease (eg, pain, dyspnea, reduced performance status). Participants who have stable disease while being treated with another agent that is not tolerated are eligible after the appropriate washout period.
   4. Dose Expansion phase ONLY:

      * Measurable disease at the time of enrollment. At least 1 measurable lesion according to RECIST v1.1 criteria. Participants must have radiographic evidence of disease progression by RECIST v1.1 criteria ≤ 6 months prior to study enrollment. Radiographic eligibility as determined by Central IUO assay.
      * Biomarker eligibility as determined by central IUO assay.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Tumor Tissue Requirements

   Dose Escalation Phase ONLY: be able to provide during Screening a tissue specimen of either a fresh biopsy of a non-target lesion or an archival tumor sample obtained within the last 6 years. A formalin-fixed paraffin-embedded (FFPE) block can be submitted or a minimum of 15 freshly sectioned unstained slides.
   1. Agree to an on-treatment biopsy to be obtained ~4-8 weeks after the initiation of REM-422 unless medically contraindicated.
   2. Dose Expansion phase ONLY: be able to provide, during Pre-Screening, a tissue specimen of either a fresh biopsy of non-targetable lesion or an archival tumor sample obtained within the last 6 years. An FFPE block can be submitted or a minimum of 15 fresh sectioned unstained slides.
6. At least 3 weeks since prior systemic non-investigational therapy at the time of start of REM- 422.
7. Toxicities from prior therapy must be stable or recovered to ≤ Grade 1. Note: Stable chronic and clinically non-significant conditions (≤ Grade 2) that are not expected to resolve are exceptions (eg, neuropathy, myalgia, alopecia, prior therapy-related endocrinopathies, etc.), and patients with these conditions may enroll.
8. Participants must be able to swallow and retain oral medications.
9. Oxygen saturation > 92% on room air or up to 2 L/min supplemental oxygen by nasal cannula with ≤ Grade 1 dyspnea.
10. Participants of childbearing potential (POCBP) must have a negative serum beta-human chorionic gonadotropin test result.
11. Participants Of Child Bearing Potential must agree to use acceptable, effective methods of contraception as outlined in Appendix 1 and not donate ova from Screening until 6 months after discontinuation of REM- 422. Women who have undergone surgical or ablative sterilization or who have been postmenopausal for ≥ 2 years are not considered to be of childbearing potential.
12. Men must agree to use acceptable, effective methods of contraception and must agree not to donate sperm from the start of receiving REM-422 until 6 months after discontinuation of REM-422.
13. Adequate bone marrow, organ function and laboratory parameters

Exclusion Criteria:

1. Known hypersensitivity or contraindication to any component of REM-422 or to drugs chemically related to REM-422 or its excipients.
2. Clinically significant active infection. Simple urinary tract infection, uncomplicated bacterial pharyngitis responding to active treatment are permitted. Participants receiving intravenous antibiotics ≤ 7 days prior to enrollment are excluded (prophylactic antibiotics, antivirals or antifungals are permitted).
3. Evidence of active HIV infection.
4. Evidence of currently active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
5. Primary immunodeficiency.
6. Current or expected need for daily systemic corticosteroid therapy ≥ 10 mg of prednisone equivalent. Topical or inhaled corticosteroids with minimal systemic absorption may enroll and continue minimal corticosteroids if the participant is on a stable dose.
7. Live vaccine ≤ 6 weeks prior to the start of REM-422.
8. Use of strong CYP3A inhibitors or CYP3A inducers
9. Drugs that reduce gastric acidity, such as H2-receptor antagonists (eg, ranitidine, famotidine) and proton pump inhibitors (e.g., omeprazole, esomeprazole) within 7 days prior to the initiation of REM-422 administration or during the study
10. Pregnancy or participants planning to become pregnant during the duration of the study, or lactation.
11. Participants with malabsorption syndrome, a disease significantly affecting gastrointestinal function, or resection of the stomach or bowel.
12. Current use of prohibited medication ≤ 1 week before starting REM-422.
13. Clinically significant cardiovascular disease:
14. Participants who have undergone major surgery (opening a mesenchymal barrier such as the pleural cavity, peritoneum, meninges, or surgical procedures requiring general anesthesia) < 4 weeks prior to enrollment.
15. History of organ transplant that requires use of immunosuppressive agents.
16. History or current autoimmune disease (eg, Crohn's disease, ulcerative colitis, rheumatoid arthritis, systemic lupus).
17. Radiation therapy ≤ 7 days prior to the start of REM-422.
18. Concurrent or previous other malignancy (other than adenoid cystic carcinoma, hematologic malignancies, or primary central nervous system [CNS] malignancies) ≤ 2 years of enrollment, except curatively treated malignancies including basal or squamous cell skin cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix.
19. Participants receiving any other investigational treatment for any indication ≤ 3 weeks prior to enrollment.
20. Unwillingness or inability to follow protocol requirements.
21. Any condition that, in the opinion of the Investigator, would interfere with evaluation of REM-422 or interpretation of the participant's safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of Treatment Emergent Adverse Events (TEAEs) | 18 months
  Frequency and severity of Treatment Emergent Adverse Events (TEAEs) will be evaluated according to the NCI-CTCAE version 5.0 and number of participants with Dose Limiting Toxicities will be assessed to determine Safety and Tolerability of REM-422
Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) | Assessed at the end of Cycle 1 for each participant
  Frequency and severity of Treatment Emergent Adverse Events (TEAEs) will be evaluated according to the NCI-CTCAE version 5.0 and the number of participants with Dose Limiting Toxicities will be assessed

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 18 months
  ORR will be evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline version 1.1 following treatment with REM-422
Median Progression Free Survival (mPFS) | 18 months
  PFS will be evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline version 1.1 following treatment with REM-422
Duration of Response (DoR) | 18 months
  DoR will be evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline version 1.1 following treatment with REM-422
Time to Response (mTTR) | 18 months
  TTR will be evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline version 1.1 following treatment with REM-422
Disease Control Rate (DCR) | 6 months
  DCR will be evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline version 1.1 following treatment with REM-422
Median Overall Survival (mOS) | 18 months
  mOS will be evaluated after treatment with REM-422
Determine pharmacokinetic profile (Cmax) of REM-422 | 18 months
  Measure Maximal concentration (Cmax) of REM-422
Determine pharmacokinetic profile (Cmin) of REM-422 | 18 months
  Measure Minimal concentration (Cmin) of REM-422
Determine pharmacokinetic profile (Tmax) of REM-422 | 18 months
  Measure Time to peak drug concentration (Tmax) of REM-422
Determine pharmacokinetic profile (AUC) of REM-422 | 18 months
  Measure Area Under the Curve (AUC) of REM-422

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bowden, MD, Study Chair — Remix Therapeutics
Locations (8):
- United States (6):
  - University of California San Francisco Helen Diller Comprehensive Cancer Center, San Francisco, California
  - Dana Farber Cancer Research Institute, Boston, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- France (2):
  - Centre Antoine Lacassagne, Nice
  - Institut de Cancerologie Gustave-Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No